CLINICAL TRIAL: NCT05108467
Title: Saving Lives by Early Detection and Treatment of Sepsis and Septic Shock by Point of Care Lactate Test in Adults
Acronym: POCLactate
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Other Study IDs: PR-21097
Record Dates: First submitted 2021-10-25; First posted 2021-11-05 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2021-11

CONDITIONS: Severe Sepsis With Septic Shock; Lactate Blood Increase
Keywords: Severe Sepsis; Septic Shock; Severe dehydration; POC Lactate; Adult
MeSH Terms: conditions — Hyperlactatemia; Sepsis; Shock, Septic; Dehydration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Case: Severe sepsis with or without shock
  Interventions: Diagnostic Test: Point of care Lactate
- Comparison: Severe dehydration with shock
  Interventions: Diagnostic Test: Point of care Lactate

INTERVENTIONS:
Diagnostic Test: Point of care Lactate — StatStrip Lactate is a handheld, point-of-care (POC) meter that brings lactate testing directly to the bedside. Lactate measured with blood gas analyzers is problematic for bedside care. Blood gas analyzers require arterial samples, large sample volumes (100-200 μL), and long analysis times (up to 2.5 minutes). In addition, blood gas analyzers are complex to use, stationary, and expensive to purchase and run.
  StatStrip Lactate testing is as easy as bedside glucose testing. Single-use, pre-calibrated biosensors provide the fastest turnaround time (13 seconds) from the smallest whole blood sample (0.6 μL) with excellent correlation to central laboratory reference methods.

SUMMARY:
Burden:

The global burden of sepsis is difficult to ascertain, although a recent scientific publication estimated that in 2017 there were 48.9 million cases and 11 million sepsis-related deaths worldwide, which accounted for almost 20% of all global deaths. Recent chart analysis from Dhaka Hospital, icddrb recorded 350 adults with severe sepsis admitted over four years. Among them, 69% of patients progressed to septic shock.

Knowledge gap:

Clinical features of shock due to sepsis and shock due to severe dehydration are very intertwining and often predicament for critical care physicians. If not recognized early and managed promptly, it can lead to septic shock, multiple organ failure, and eventually death. Serum lactate may play a role as the point of care test in differentiating shock due to severe sepsis from shock due to severe dehydration.

Relevance:

Being the largest diarrhoeal disease hospital, the Dhaka Hospital of icddr,b is ideal for researching shock with diarrheal diseases. Even though the onset of sepsis can be acute and poses a short-term mortality burden, it can also cause significant long-term morbidity, requiring treatment and support. Thus, addressing sepsis and severe sepsis by early detection and prompt management should be a comprehensive way to reduce the burden in our community.

DETAILED DESCRIPTION:
The global burden of sepsis is difficult to ascertain, although a recent scientific publication estimated that in 2017 there were 48.9 million cases and 11 million sepsis-related deaths worldwide, which accounted for almost 20% of all global deaths. Recent chart analysis from Dhaka Hospital recorded 350 adults with severe sepsis admitted to a diarrheal hospital over four years, among them, 69% of patients progressed to septic shock.

If not recognized early and managed promptly, it can lead to septic shock, multiple organ failure, and death. It is most frequently a serious complication of infection, particularly in low- and middle-income countries. Early diagnosis and timely and appropriate clinical management of sepsis, such as optimal antimicrobial use and fluid resuscitation, are crucial to increase the likelihood of survival. Even though the onset of sepsis can be acute and poses a short-term mortality burden, it can also be the cause of significant long-term morbidity requiring treatment and support. Thus, sepsis requires a multidisciplinary approach.

Shock may occur as a ramification of severe sepsis, and on the other hand, a patient may present with shock due to severe dehydration from severe diarrhea. However, the differentiation of shock as a cascade of severe sepsis from the shock due to severe dehydration is intriguing. Fluid management in these two entities is different, although the initial bolus (30 ml/kg) in both cases is the same. If fluid management could not be done efficiently, some patients might end up with fluid overload especially in case of shock due to severe sepsis and under hydration in case of shock due to severe dehydration. On the other hand, there could be also overuse of inotropes if we are unable to identify the requirement of additional fluid. Thus, we need to have a point of care biomarker that may guide us further fluid requirement (or requirement of inotrope) after the initial bolus. Not only is severe sepsis the most common non-cardiac cause for intensive care unit (ICU) use, it has emerged as a major driver of hospital costs in developing countries.

Serum lactate level, which measures the level of lactic acid in the blood, is a fairly reliable and accurate indication of tissue hypoperfusion and hypoxia. The signs and symptoms, which may vary from patient to patient, include altered mental status; pale, cool, clammy skin; nausea and vomiting; diaphoresis; hypotension; tachypnea; and tachycardia. Surprisingly all these features are evident in severe sepsis or severe dehydration. In addition, septic shock is often associated with macrocirculatory dysfunction causing arterial hypotension, microcirculatory dysfunction, and decreased oxygen and nutrient extraction by peripheral tissues. Thus, lactic acid levels have become a useful marker for tissue hypoperfusion and may also serve as an endpoint for resuscitation in patients with sepsis and septic shock.

Serum lactate is proven to be an ideal point of care test to diagnose severe sepsis or septic shock successfully. On the other hand, although there is very limited knowledge regarding the utility of serum lactate in severe dehydration, evidence showed a reduction of serum lactate level after successful hydration.

Based on this evidence, we aimed to conduct this prospective exploratory study of serum lactate to differentiate severe dehydration from severe sepsis.

Methodology:

Study design: This is an observational exploratory study to find out the role of serum lactate to differentiate patients having shock due to severe sepsis and shock due to severe dehydration.

Primary Objectives:

Role of serum lactate to identify the requirement of inotropes between patients having shock due to severe sepsis and shock due to severe dehydration.

Secondary Objectives:

i) Prognostic accuracy of serum lactate level for mortality outcome among adults with severe sepsis or septic shock.

ii) Prevalence of severe sepsis or septic shock among diarrheal patients.

Study duration:

12 months (Patient enrolment will be continued for completed six months)

Sample Size Calculation This will be an eight months' time-bound study. In the last six months in 2021, we have evaluated 198 patients in our suspected COVID-19 tent, where 78 were suspected of severe sepsis or septic shock. Based on this assumption we expect to enroll consecutive 80 patients, each with severe sepsis and/or shock, and 80 patients with only severe dehydration without any other associated co-morbidities.

Data analysis Data will be analyzed by using SPSS, STATA and Epi info by the investigators and statisticians of icddr,b. The primary endpoint of this trial is the difference of serum lactate levels in shock due to severe sepsis group and shock due to severe dehydration group. For comparison of parametric continuous variable, we will use paired t-test. For non-parametric continuous variable, we will use Mann Whitney U test. For comparison of the dichotomous or categorical variables such as: requirement of multiple inotropes, duration of hospitalization, mortality during hospitalization and bacterial isolation from blood or stool we will use Chi square test and the Fisher's exact test if the expected frequency of any cell is less than 5.

Odds ratio (OR) and their 95% confidence intervals (CIs) were used to demonstrate the strength of association. For statistically significant, a p-value is set <0.05. To identify association of high lactate level with severe sepsis in diarrheal adults, initially, a bivariate model will be built, and then a multivariable regression analysis model identified factors independently associated with severe sepsis after controlling for the relevant confounding variables.

ELIGIBILITY:
Inclusion Criteria:

* Patients have shock due to severe sepsis or septic shock.
* Consent to participate in the study from the patient or his accompanying caregiver.

Exclusion Criteria:

* Any emergency which might require urgent referral within half an hour of admission.
* Known case of cancer or chemotherapy.
* Life-threatening conditions required cardiopulmonary resuscitation (CPR) on arrival.
* Cardiac shock or anaphylactic origin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diarrhea is the entry point for admission to the hospital. Adults presenting with diarrhea and clinically defined and severe sepsis or septic shock recommended by surviving sepsis guidelines supported with our local evidence will be selected as participants in the study. Adults presenting with severe dehydration assessed by the admitting doctor will be enrolled as a comparison group for comparing the role of lactate in both conditions.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-10-21 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in serum lactate level after completion of hydration in the presence of clinical features of severe sepsis and shock | Within 90 minutes of enrollment
  First sample (POC-1): Lactate level on enrolment Second sample (POC-2): Lactate level after fluid bolus Expected outcome: Change in level of POC Lactate will be significant in those who do not require inotropes compared to those who require inotropes.

SECONDARY OUTCOMES:
Requirement of multiple inotropes | Within 6 hours of enrollment
  Through looking at the POC lactate test, prediction of requirement of more than one ionotrops

CONTACTS AND LOCATIONS:
Locations (1):
- International Centre for Diarrheal Disease Research, Bangladesh, Dhaka, Outside U.S. and Canada, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
The full data is accessible as per the data sharing policy of icddrb through Research Administration.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the publication of research findings in peer reviewer journal
Access Criteria: Communication with the Research Administration of icddrb through the website
URL: http://shetu.icddrb.org/ra-overview

REFERENCES:
- [Derived] Shahrin L, Sarmin M, Parvin I, Al Hasan MM, Nahar MA, Mohammad Sayeem Bin Shahid AS, Shaima SN, Salahuddin Mamun GM, Nasrin S, Ahmed T, Chisti MJ. Point of care lactate for differentiating septic shock from hypovolemic shock in non-ICU settings: a prospective observational study. Lancet Reg Health Southeast Asia. 2024 Oct 21;30:100500. doi: 10.1016/j.lansea.2024.100500. eCollection 2024 Nov. PMID 39502270